CLINICAL TRIAL: NCT01744899
Title: The Influence of Different Sitting Postures on Soleus H-Reflex in Normal Subjects
Brief Title: Soleus H-Reflex in Different Sitting Postures
Status: Completed | Type: Observational
Sponsor: Texas Woman's University (Other)
Collaborators: The Saudi Arabian Cultural Mission to the United States (Unknown)
Responsible Party: Principal Investigator, Hamad Al Amer, Mr, Texas Woman's University
Other Study IDs: 16518
Record Dates: First submitted 2012-09-26; First posted 2012-12-07 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Compression of Spinal Nerve Root; Spinal Disorder; Low Back Pain
Keywords: Lumbosacral spine; Nerve roots; Sitting; H-reflex
MeSH Terms: conditions — Radiculopathy; Spinal Diseases; Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Prolonged sitting: Includes individuals who spent an average of at least 6 hours a day sitting over the past year.
  Interventions: Other: Sitting posture
- Control: Includes individuals who spent 4 hours or less/day sitting over the past year.
  Interventions: Other: Sitting posture

INTERVENTIONS:
Other: Sitting posture — The outcomes were measured while the participants assumed erect, slumped and slouched sitting postures.

SUMMARY:
The purpose of this study was to examine the effect of prolonged sitting duration and three different sitting postures (erect, slumped, and slouched sitting postures) on spinal nerve root function by measuring the soleus (SOL) H-reflex amplitude. In addition, the pressure under the ischial tuberosities during the three sitting postures were assessed and correlated with the SOL H-reflex amplitude.

DETAILED DESCRIPTION:
Participants were assigned to two groups (prolonged sitting group and controls) based on their daily sitting duration with 15 participants in each group. The outcome measures were recorded during erect, slumped and slouched sitting postures. The differences between the two groups and the three sitting postures in the outcome measures were examined for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, speak, and understand English

Exclusion Criteria:

1. Current complaint of low back pain.
2. Current injury to the ankle and/or foot.
3. Limited ankle movement.
4. Leg length discrepancy.
5. Scoliosis.
6. History of:

   * Back surgery.
   * Calf muscle injury/surgery.
   * Radicular symptoms.
   * Peripheral neuropathy.
   * Upper motor neuron lesion.
   * Systemic and metabolic diseases.
   * Cancer.
7. Pregnant at the time of the study.
8. Use of pain medications at the time of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults from both genders.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Lumbosacral nerve root function by as measured by the soleus H-reflex amplitude | The outcome was measured during one session that lasted for an average of 3 hours. No further measurement was performed after that session.

SECONDARY OUTCOMES:
Pressure under the ischial tuberosities | The outcome was measured during one session that lasted for an average of 3 hours. No further measurement was performed after that session.
  Pressure under the ischial tuberosities was measured in millimeter of mercury (mmHg), with 0 mmHg representing no ischial pressure and 644 mmHg representing the highest pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Hamad S Al Amer, MS, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's University, Houston, Texas, United States